CLINICAL TRIAL: NCT03944343
Title: Validation of a New Antidiabetic Food Concept Based on the Modulation of the Intestinal Flora
Brief Title: Prebiotic Effects on Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, senior lecturer, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/1
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Diet Prevention of Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized crossover study design. Healthy young adult volunteers.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Reference product (Sham Comparator): Commercial cereals and a commercial yogurt
  Interventions: Other: Cereal based products
- Test product A (Experimental): Specific designed cereals A and yogurt
  Interventions: Other: Cereal based products
- Test product B (Experimental): Specific designed cereals B and yogurt
  Interventions: Other: Cereal based products
- Test product C (Experimental): Specific designed cereals C and yogurt
  Interventions: Other: Cereal based products
- Test product D (Experimental): Specific designed cereals D and yogurt
  Interventions: Other: Cereal based products

INTERVENTIONS:
Other: Cereal based products — The cereal products are made from common Swedish cereals.

SUMMARY:
The primary purpose of this project is to evaluate effects in healthy humans on glucose tolerance of cereal products with high amounts of fermentable dietary fibre. Secondary issues are to investigate effects of the test foods on subjective appetite variables, mood variables and gut microbiota composition. The test food products will be consumed in the evening and test variables will be determined the next morning. The study will apply a randomized crossover study design.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2
* age 20-40 years
* normal diet
* healthy

Exclusion Criteria:

* fasting blood glucose >6.1
* diagnosed or known disease
* known gastrointestinal disorder
* food allergies or intolerance
* special diet regiments
* smokers

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 3 hours
  The incremental (3 hours) blood glucose area under the curve after a standardized breakfast, following consumption of the test- or reference products the previous evening. Glucose concentrations will be analysed from capillary blood at fasting and at 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min and 180 min after the standardized breakfast.

SECONDARY OUTCOMES:
Subjective appetite variables | 3 hours
  Determination of appetite variables (satiety, hunger and desire to eat) at fasting in the morning and after the standardized breakfast following consumption of the test- or reference products the previous evening. The appetite sensations will be determined at fasting and then at 30 min, 60 min, 90 min, 120 min, 150 min and at 180 min. The variables will be determined by registration on a 0-100 mm visual analogue scales (VAS). Higher ratings are considered to be better for the rating of satiety meanwhile lower ratings are considered to be better for hunger and desire to eat.
Mood parameters | 3 hours
  Determination of mood variables (activity and valence) at fasting in the morning and after the andardized breakfast, following consumption of the test- or reference products the previous evening. The mood variables will be determined at fasting and then at 60 min, 120 min and at 180 min. The variables will be determined by registration on a 0-100 mm visual analogue scales (VAS).
Breath hydrogen | 3 hours
  Determination of breath hydrogen concentrations will be performed at fasting and after the standardized breakfast, following consumption of the test- or reference products the previous evening. Breath hydrogen will be determined at fasting and then at 30 min, 60 min, 90 min, 120 min, 150 min and at 180 min. Breath hydrogen will be measured by exhaling in a portable measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, associate professor, Principal Investigator — Lund University
Locations (1):
- Lund University, Food Technology, Engineering and Nutrition, Lund, Sweden